CLINICAL TRIAL: NCT02037932
Title: Hydrogel Balloon Assisted Intracranial Aneurysm Coiling Registry
Acronym: GELATIN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00021229
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Intracranial Aneurysms; Aneurysm; Brain Aneurysm
Keywords: Aneurysm; Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon Assisted Coiling (Experimental): Balloon Assisted Coiling using MicroVention second-generation hydrogel coils and MicroVention Scepter Occlusion Balloon Catheter.
  Interventions: Device: Balloon Assisted Coiling using MicroVention second-generation hydrogel coils and MicroVention Scepter Occlusion Balloon Catheter.

INTERVENTIONS:
Device: Balloon Assisted Coiling using MicroVention second-generation hydrogel coils and MicroVention Scepter Occlusion Balloon Catheter. — Balloon Assisted Coiling using MicroVention second-generation hydrogel coils and MicroVention Scepter Occlusion Balloon Catheter.
  Other Names: MicroVention hydrogel coils; MicroVention Scepter C; MicroVention Scepter XC

SUMMARY:
The objective of the GELATIN registry is to prospectively evaluate intracranial aneurysm occlusion and retreatment rates as well as adverse event rates in patients undergoing balloon-assisted coiling using the MicroVention Scepter Occlusion Balloon Catheter and second-generation MicroVention hydrogel coils for treatment of previously treated or untreated ruptured and unruptured intracranial aneurysms.

DETAILED DESCRIPTION:
This is a prospective, single arm, single center study of patients with ruptured or unruptured saccular aneurysms that are embolized using MicroVention second-generation hydrogel coils and undergo balloon remodeling with the MicroVention Scepter Occlusion Balloon Catheter. Data for each patient will be collected 6 ± 3 months post-procedure for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-80 years of age.
* Patient has a documented, previously treated or untreated saccular intracranial aneurysm, 4- 20 mm unruptured or ruptured, suitable for treatment with balloon assisted coil embolization.
* Target aneurysm has a neck ≥4mm or the largest diameter to neck ratio of 2 or less.
* Patient has a Hunt and Hess Score of 3 or less.
* Patient has a premorbid mRS of 3 or less.
* Patient or patient's legally authorized representative has provided written informed consent.
* Patient is willing to and can comply with study follow-up requirements.

Exclusion Criteria:

* Inability to obtain informed consent.
* Patient is <18 or >80 years of age.
* Target aneurysm is dissecting, fusiform, mycotic, or arteriovenous malformation-related.
* Aneurysm that was treated previously with stent-assisted coiling.
* Implantation of the stent after the balloon-assisted coiling or combined stent and balloon assisted coiling.
* Target aneurysm is deemed unsuitable for balloon-assisted coiling by the treating physician prior to the procedure.
* Target aneurysm will be treated with a total coil length comprised of less than 80% second generation MicroVention Hydrogel Coils.
* Balloon-assisted coiling will be performed using a balloon catheter other than the MicroVention Scepter balloon (Scepter C, Scepter XC, any future Scepter configurations).
* Patients in which the target aneurysm is planned not to be coiled in one procedure (i.e. staged procedure).
* Patients with more than one aneurysm that requires treatment. (However, a second small low risk aneurysm that does not require therapy may be allowed.)
* Patients with a life expectancy of ≤ 9 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Aneurysm recurrence rate | 3-9 month follow-up

SECONDARY OUTCOMES:
Occlusion Rate | At immediate post-procedure (Day 1) and 3-9 month follow-up
  Angiographic occlusion of the aneurysm will be adjudicated using immediate post-procedure and 3-9 month follow-up angiography.
Number of coils used | At end of study procedure (Day 1)
Total coil length used | At immediate post-procedure (Day 1)
Aneurysm re-treatment rate | 3-9 month follow-up
Aneurysm Bleed and Re-bleed Rate | 3-9 month follow-up
  Aneurysm Bleed and Re-bleed Rate will be assessed and recorded at the 3-9 month follow-up.
Time of fluoroscopic exposure | At immediate post-procedure (Day 1)
  Total time of fluoroscopic exposure will be captured from the initial recording of the road map to the final angiogram after completion of the coil embolization procedure.
Modified Rankin Score | At baseline (Day 1) and hospital discharge (Day 3) and 3-9 month follow-up
  Modified Rankin score will be recorded at baseline, hospital discharge, and during the 3-9 month follow-up.
Device-related serious adverse events | From the study procedure (Day 1) until 3-9 month follow up
  Procedural and post-procedural serious adverse events related to the device and/or procedure will be captured and recorded at the end of the procedure and until the patient has completed the 3-9 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Osama O Zaidat, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States